CLINICAL TRIAL: NCT05549063
Title: Effect of Different Exercise Approaches on Balance and Proprioception in Individuals With Pes Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pes planus
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pes Planus
Keywords: Exercise; Stability exercises; Mobility exercises; Stretching exercises
MeSH Terms: conditions — Flatfoot; Motor Activity | interventions — Range of Motion, Articular; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: It is planned to randomly divide 40 individuals diagnosed with pes planus by the physician into two.
  In these groups, there should be a pes planus problem on both sides. The first group will be given stretching exercises, while the second group will be given mobility and stability exercises.
Who Masked: Participant, Investigator
Masking Description: Evaluation and treatment will be carried out by different physiotherapists. In this way, it is aimed to provide an objective evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobility and Stability Exercise (Experimental): The patients were divided into two groups. Exercises were applied to both groups for 4 weeks.
  Interventions: Other: Mobility and Stability Exercise
- Stretching Exercise (Active Comparator): The patients were divided into two groups. Exercises were applied to both groups for 4 weeks.
  Interventions: Other: Stretching Exercise

INTERVENTIONS:
Other: Mobility and Stability Exercise — Mobility and stability exercises
  Arms: Mobility and Stability Exercise
Other: Stretching Exercise — Balance and reaching exercise
  Arms: Stretching Exercise

SUMMARY:
Pes planus; It can be defined as the valgus of the hindfoot while loading the foot, the disappearance of the medial longitudinal arch in the midfoot, and the supination of the forefoot relative to the hindfoot. It may also occur due to the fact that the medial longitudinal arch in the foot is lower than the required height according to the anatomical position. The parts of the foot that touch the ground are anatomically healthy in a person; They are the heads of the calcaneus tuberositas calcanei on the back of the foot and the 5 metatarsal bones on the front of the foot. In the standing position, 25% of our body weight is on the tuber calcanei, while 25% is on the 5 metatarsal bones. In individuals with pes planus, convergence of the sole of the midfoot to the ground may even result in the sole of the midfoot touching the ground at its advanced levels. It is one of the common foot deformities.

DETAILED DESCRIPTION:
Pes planus can cause symptoms and dysfunction that are symptomatic or severe enough to limit patients' quality of life. Degeneration of the posterior tibial tendon may occur due to trauma, neuroarthropathy, neuromuscular disease and inflammatory arthritis. Among these, the most common cause of pes planus is the degeneration of the posterior tibial tendon.

The highest arch of the foot, the medical longitudinal arch calcaneus, talus, navicular, cuneiform and 1-2-3. It is formed by metatarsals. It is effective in the distribution of the load on the feet. Plantar ligaments are important in protecting the dome of the foot.

They used many definitions known as pes planus, that is, flat feet in the literature. Weak foot, relaxed foot, pes valgus, congenital hypermobile flat foot, hypermobile flat foot, flaccid flat food, talipes calcaneovalgus, compensated talipes equinus can be given as examples.

Balance disorders and general joint hypermobility are among the clinical symptoms of pes planus. In a study conducted with 100 individuals aged between 18 and 45, when the balance time of individuals without pes planus was compared with the balance time of individuals with pes planus; It was determined that individuals without pes planus had better balance times. It has been determined that as the degree of pes planus increases, the time to stay in balance decreases in individuals.

Stretching exercises; It is defined as the pulling force applied to lengthen the muscle and connective tissues in the human body. Stretching exercises are divided into 4 in themselves. These; dynamic stretching, static stretching, ballistic stretching and PNF stretching.

Mobility exercises; It consists of low-speed, variable-intensity, repetitive, passive movements applied to joints and ligaments within the normal range of joint motion.

Stability exercises; It is defined as the ability to control joint movement or position by coordinating the movements of the surrounding tissues and neuromuscular system.

ELIGIBILITY:
Inclusion Criteria:

* Having mild and moderate pes planus,
* Volunteering of individuals,
* Being between the age group of 18-40,
* Having experienced at least one inflammatory symptom (pain, swelling, etc.)
* Not having any systemic, locomotor and foot related diseases, sensory loss, diabetic and peripheral neuropathy.

Exclusion Criteria:

* Having had a serious lower extremity injury in the last 6 months,
* Getting a full score from the balance test,
* Having ligament rupture in the ankle.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-17 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Star Excursion Balance Test | 4 weeks
  It is used to measure dynamic postural balance. The test is based on the ability to reach the farthest possible distance on the supporting leg in 8 different directions.
  The person reaches as far as he can reach with his foot and touches the strip lightly with the tip of his toe. Then it returns to the starting position. Then the other line is passed and a total of 8 lines are completed in this way. After the whole process is repeated 3 times with the right foot, the left foot is changed and it is repeated 3 times. The participant records the distances reached at the end of the test. We have 16 scores left for 8 right and 8 left feet in total.
  Reach (%) = Reach distance / Leg length x 100
Range of Motion Measurement | 4 weeks
  Dorsiflexion, plantar flexion, inversion and eversion ranges of motion of the ankle joints of individuals are actively measured using a universal goniometer and recorded in degrees.
Berg Balance Test | 4 weeks
  Berg Balance Test It consists of 14 general balance activities that change the orientation of the body's center of gravity with respect to the support surface and evaluate the ability to maintain a static position while decreasing on the support surface. During the activities, the patient is evaluated by the observer, and the score for each activity is determined, ranging from 0 to 4. The highest score corresponds to the ability to complete the activity quickly and easily. The highest overall score is 56 and reflects a perfect balance function. The closer the score is from 56 to 36, the greater the risk of falling. It is described as a 'gold standard' test in functional balance evaluation.
Weight-bearing Lunge Test Weight-bearing lunge test | 4 weeks
  Dorsi flexion range of motion was measured as the range of motion of the ankle joint. In the test, the patient was initially positioned standing against the wall. The second toe and heel of the foot to be measured were adjusted so that the midpoint of the knee was perpendicular to the wall. Then, the patient was asked to move forward without lifting his heel off the ground, and to touch his knee to the wall. The furthest distance that the patient could touch the wall without raising the heel was determined. The distance between the tip of the second finger and the wall was measured in cm. Three trials were performed and the mean value was recorded for analysis. Test is a valid and reliable test for measuring dorsiflexion.

SECONDARY OUTCOMES:
Functional Reach Test | 4 weeks
  The results do not adequately represent functional activities in daily life, since in many test protocols for evaluating the stability limits of the individual, the evaluation is performed during forward bending without using the upper extremity.
  Functional reach is a function that takes place in many daily activities and creates constant stress on balance. Voluntary upper extremity movements are accompanied by postural stabilizing activities of the leg and trunk muscles, and postural control mechanisms must be preserved for upper extremity movements in the standing position.
  It is defined as the maximum distance that an individual can reach forward in the horizontal plane while maintaining stability on the support surface in the standing position.
  Functional reach; It can be measured in two ways as electronic functional reach measurement and functional reach measurement with tape measure.
  Measuring with a tape measure is very practical.
Manual Muscle Test | 4 weeks
  Manual Muscle Test, which scored individuals' muscle strength values between 0 and 5, was used. In the muscle test, the patient is placed in the starting position of the movement and asked to do the movement. Motivation is increased by giving verbal warnings.
  Muscle tests should be started with a value of 3. If the patient can easily make this value, the values of 3+, 4 and 5 are checked. If it cannot reach the value of 3, the values of 2.1 and 0 should be checked.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçeşehir University, Istanbul, Turkey (Türkiye)